CLINICAL TRIAL: NCT00505986
Title: Genomic Endometrial Expression in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Jose Bellver, Gynecologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: VLC-JB-0507-607-29
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Obesity and Embryo Implantation
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Procedure: endometrial biopsy

SUMMARY:
Determine if different genomic endometrial expression exists during embryo implantation in obese women in comparison with non obese women.

ELIGIBILITY:
Inclusion Criteria:

* group A: non obese oocyte donors (BMI: 18 - 29 kg. /m2)with proven fertility
* group B: obese oocyte donors: (BMI: >29 kg./m2)with proven fertility
* group C: obese (BMI: >29 kg./m2) infertile patients,

Exclusion Criteria:

* recurrent miscarriage

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Bellver, MD PhD, Principal Investigator — Instituto Valenciano de Infertilidad
Locations (1):
- Instituto Valenciano de Infertilidad Spain, Valencia, Valencia, Spain